CLINICAL TRIAL: NCT01182363
Title: Reducing Risk After an Adverse Pregnancy Outcome: Addressing Maternal Depression During Internatal Periods
Brief Title: Reducing Risk After an Adverse Pregnancy Outcome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H28906
Record Dates: First submitted 2010-07-28; First posted 2010-08-16 (Estimated); Last update posted 2014-08-28 (Estimated); Status verified 2014-08

CONDITIONS: Maternal Depression
Keywords: maternal depression; prematurity; early intervention; developmental delay
MeSH Terms: conditions — Premature Birth; Learning Disabilities

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention): Usual early intervention services
- Problem Solving Education (Experimental)
  Interventions: Behavioral: Project Solve Education

INTERVENTIONS:
Behavioral: Project Solve Education — Problem solving education (PSE), a brief skills-building psychotherapeutic intervention that focuses on specific daily problems, and applies to these problems a structured approach to finding and evaluating solutions, is one such problem solving approach. Problem solving education differs from other problem solving interventions in that it can be conducted by a variety of health providers, who do not have specific training as mental health clinicians. Sessions are fairly brief (approximately 30 minutes in length) and positive, sustained effects have been achieved in 6-8 sessions. Problem solving education's success is based on premise that strong problem solving abilities promote a sense of control and self-efficacy and buffer the negative effects of life stressors.
  Arms: Problem Solving Education

SUMMARY:
This application to the Boston University Medical Center Institutional Review Board outlines a research plan devoted to identifying and managing maternal depression in Early Intervention (EI). The target population is women who's children are enrolled in early intervention who have experienced an adverse pregnancy outcome, defined as the birth of a child who was born prematurely, low birth weight, or with birth defects. Early intervention provides developmental services to the state's birth to three population under the Part C of the Individuals with Disabilities Act (IDEA). Our intervention strategy involves the identification of mothers whose children receive early intervention services and who, themselves, are at risk for depression. Eligible mothers will be offered a preventative intervention that involves the principles of Problem Solving Treatment (PST). Problem Solving Treatment is a brief skills-building psychotherapeutic intervention that focuses on specific daily problems, and applies to these problems a structured approach to finding and evaluating solutions.

This study will be a parallel group randomized control trial (RCT) of 188 mother-child dyads. Mothers in the intervention group will receive 6 sessions of Problem Solving Treatment, which will be referred to as Problem Solving Education (PSE) in this application. The women in the control site will receive usual care. Problem Solving Education interventionists (Problem Solving Educators or PS Educators) will conduct Problem Solving Education with mothers of children who receive early intervention services through Thom Child and Family Services, Bay Cove Early Intervention program, South Shore Mental Health (Step One Early Intervention), and Meeting Street Early Intervention with an enrollment goal of 188 mothers. In addition to engaging in Problem Solving Education sessions, mothers who agree to participate in the study will meet with research staff to complete 1)baseline assessment measures at study enrollment and 2) outcome assessment measures 3 months after baseline assessment and 3) outcome assessment measures 6 months after baseline assessment.

DETAILED DESCRIPTION:
Community-based programs that target vulnerable families consistently identify maternal depression as a factor that negatively impacts maternal and child outcomes. A population in particular need of mental health interventions are mothers of children with who have experienced an adverse pregnancy outcome, defined as the birth of a child who was born prematurely, low birth weight, or with birth defects, a group with increased incidence of depression. Children of depressed mothers are at risk for a vast range of poor physical, cognitive, and emotional problems. Children who have existing underlying developmental concerns due to adverse birth circumstances are especially vulnerable. Therefore, identifying at-risk mothers and intervening to prevent the onset or re-occurrence of depression represents an opportunity not only to help the women affected, but also to improve developmental and behavioral outcomes for their children. Children under 3 with conditions that impact their developmental trajectories receive services through federally mandated Early Intervention (EI) programs; thus early intervention is an important, but underutilized, setting for identification and intervention with at-risk mothers. While effective preventative psychosocial treatments for depression exist, none have been delivered and evaluated in the context of a home-based program specifically for mothers of infants and children with developmental and other chronic health conditions.

The demographics of early intervention families suggest that mothers of enrolled children are at risk for depressive illness. Families are poorer (1 in 4 received welfare payments in the past year), mothers less well educated, and African-Americans are overrepresented (21% vs. 14% of general population), reflecting known risk factors for depression. Almost half of the infants who enter early intervention in the first year of life, the target group for the proposed intervention, are low birth weight (LBW) and have significantly higher levels of demographic risk factors than their normal birth weight peers. Numerous studies have documented elevated incidence of depression among mothers of early born infants. The youngest early intervention enrollees are also more likely to have identified disabilities or conditions, such as cerebral palsy and requirements for assistive technologies that have also been associated with higher rates of maternal depressive symptoms

Strong problem-solving abilities serve as important buffers against the negative impact of life stressors; whereas limited problem solving skills have been linked to the cause and persistence of psychological disorders. Problem solving approaches to depression prevention and treatment are rooted in research that has demonstrated that minor life events or problems are highly correlated with psychological distress, in general, and with depression, specifically. Problem solving interventions that promote skill building have demonstrated effectiveness in reducing behavioral risk, including depression, in a number of settings. Problem solving education (PSE), a brief skills-building psychotherapeutic intervention that focuses on specific daily problems, and applies to these problems a structured approach to finding and evaluating solutions, is one such problem solving approach. Problem solving education differs from other problem solving interventions in that it can be conducted by a variety of health providers, who do not have specific training as mental health clinicians. Sessions are fairly brief (approximately 30 minutes in length) and positive, sustained effects have been achieved in 6-8 sessions. Problem solving education's success is based on premise that strong problem solving abilities promote a sense of control and self-efficacy and buffer the negative effects of life stressors.

The effectiveness of Problem solving education has been well documented in reducing depressive symptoms and increasing function among patients with major depression and possibly minor depression and dysthymia. We propose a research plan that involves delivering Problem solving education to at risk mothers to (i) directly reduce symptom burden among mothers with depressive symptoms, and (ii) facilitate access to further mental health services.

ELIGIBILITY:
Inclusion Criteria:

* Mothers of children with a child < or equal to 18 months of age
* Mothers who speaks English or Spanish
* Mothers of children who receive early intervention services for a condition related to an adverse pregnancy outcome (gestational age less than 37 weeks, birth weight less than 2500 grams, congenital, genetic or other condition expected to result in chronic health condition or developmental delay, Neonatal Intensive Care Unit admission great than 5 days, Apgar of 5 at 5 minutes).
* Mother meets depression risk criteria in 2/4 areas of risk (current depressive symptoms, risk factors for depressive illness, social risk, limited financial resources).

Exclusion Criteria:

* Women whose children are not currently enrolled in early intervention.
* Lack capacity to understand study procedures and provide consent
* Plan to relocate to another geographic region within 6 months
* Current psychosis
* Active suicidal ideation
* Diagnosis of schizophrenia.
* Mother actively using illicit drugs.
* Child's adverse birth outcome is not expected to result in chronic health condition or developmental delay.

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 188 (Actual)
Dates: Start 2010-08; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Quick Inventory of Depressive Symptomology | Baseline

SECONDARY OUTCOMES:
Parent Stress Index | Baseline
Social Adjustment Scale - Self-report (SAS- SR) | Baseline
Perceived Stress Scale | Baseline
Social Problem Solving Inventory | Baseline

CONTACTS AND LOCATIONS:
Overall Officials: Emily Feinberg, ScD CPNP, Principal Investigator — Boston University
Locations (4):
- United States (4):
  - Bay Cove Early Intervention, Boston, Massachusetts
  - THOM Child and Family Services, Natick, Massachusetts
  - South Shore Mental Health Step One Early Intervention, Quincy, Massachusetts
  - Meeting Street, Providence, Rhode Island